CLINICAL TRIAL: NCT04842487
Title: Lenalidomide Combined With Anti-CD20 Monoclonal Antibodies-CHOP in Untreated Diffuse Large B-Cell Lymphoma Patients With MYC and BCL2 Co-expression : An Open-lable，Multicenter，Phase II Study
Brief Title: R2-CHOP in Untreated DEL-DLBCL：An Open-lable，Multicenter，Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-052-01
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2020-06

CONDITIONS: DLBCL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): 1. Lenalidomide：25mg po QN,D1-10
  2. Rituximab: 375mg/m2, ivdrip, D1
  3. CTX: 750mg/m2, iv or ivdrip, D1
  4. THP: 50mg/m2, iv or ivdrip, D1
  5. VCR： 1.4 mg/m2 , iv（max：2mg）, D1
  6. Pred: 60mg/m2, po, D1-5
  Interventions: Drug: R2-CHOP(Lenalidomide,Rituximab,cyclophosphamide，hydroxyldaunorubicin，Vincristine，Prednisone）)

INTERVENTIONS:
Drug: R2-CHOP(Lenalidomide,Rituximab,cyclophosphamide，hydroxyldaunorubicin，Vincristine，Prednisone）) — Lenalidomide：25mg po QN,d1-10 Rituximab: 375mg/m2, ivdrip, d1 Cyclophosphamide: 750mg/m2, iv or ivdrip, d1 Hydroxyldaunorubicin: 50mg/m2, iv or ivdrip, d1 Vincristine： 1.4 mg/m2 , iv（max：2mg）, d1 Prednisone: 60mg/m2, po, d1-5 every 3 weeks was a course of treatment

SUMMARY:
To assess the efficacy and safety of lenalidomide combined with rituximab, vincristine, doxorubicin, cyclophosphamide, and prednisone (r2-chop) in the initial treatment of DEL-DLBCL. The primary endpoint is the complete response rate, and the second endpoints are survival time (OS and PFS) and overall response rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MYC and BCL2 co-expression Diffuse Large B-Cell Lymphoma diagnosed by histopathologyImmunohistochemistry confirmed that the positive expression rate of BCL-2≥50% and c-Myc≥ 40%.
* Male or female patients: 18-80 years old.
* ECOG physical condition score: 0-2 points for patients.
* IPI score≥3.
* Patients have not received any anti-tumor therapy such as radiotherapy, chemotherapy, targeted therapy or stem cell transplantation.
* In those patients with at least one evaluable or measurable lesion meeting Lugano 2014 criteria, the evaluable lesion was: 18F fluorodeoxyglucose / positron emission tomography (18FDG / PET) examination showed that the uptake of lymph nodes or extranodal areas was increased (higher than that of liver) and pet and / or computed The features of tomography (CT) were in accordance with lymphoma. The measurable lesions were nodal lesions with a length of > 15 mm or extranodal lesions with a length of > 10 mm, accompanied by an increase in 18FDG uptake. There was no measurable lesion and the uptake of 18FDG was increased.
* Patients with good function of main organs, i.e. one week before admission, met the following requirements: WBC >= 3.5×10^9 / L, NEU≥1.5×10^9/L, Hb >= 80g / L, PLT >= 100 ×10^9 / L; heart and liver functions were normal (total bilirubin <= 1.5 times of normal value, ALT and AST <= 2.5 times of normal value), renal functions were normal (serum creatinine <= 1.5 times of normal value), and coagulation function was not abnormal.
* LVEF≥50%, measured by echocardiography.
* No other tumor-specific concomitant therapy has been administered (including steroids).
* Pregnant women of childbearing age must have a pregnancy test (serum or urine) within 14 days before enrollment and the result is negative, and they are willing to use reliable methods of contraception during the test.
* Patients have no other serious diseases in conflict with this clinical trial protocols.
* The subjects who volunteer to join the study and sign the informed consent form, have good compliance and cooperate with the follow-up.

Exclusion Criteria:

* Other types of DLBCL: Diffuse large B-cell lymphoma associated with chronic inflammation, lymphomatoid granulomatosis, Primary mediastinal (thymic) large B-cell lymphoma, ALK-positive large B-cell lymphoma, Primary effusion lymphoma, Burkitt lymphoma, High-grade B-cell lymphoma(including High-grade B-cell lymphoma, NOS, High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements), B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classic Hodgkin lymphoma, Primary diffuse large B-cell lymphoma of the CNS, EBV-positive diffuse large B-cell lymphoma.
* Transformed DLBCL (transformed DLBCL from follicular lymphoma, chronic lymphocytic leukemia/small B lymphocytic lymphoma), Diffuse large B-cell lymphoma with secondary involvement of the central nervous system (SCNS-DLBCL).
* Other malignancies within the past 5 years except for carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Major surgical procedures (excluding diagnostic surgical procedures) performed in the past 2 months.
* Prior treatment for NHL, concomitant chemotherapy, radiotherapy immunotherapy, monoclonal antibody therapy, surgical treatment (except for diagnostic surgery and biopsy).
* Prior treatment with cytotoxic drugs or anti-CD20 monoclonal antibody for other conditions (e.g. Rheumatoid arthritis)
* Prior treatment with thalidomide, lenalidomide, or other drugs.
* Prior treatment with any monoclonal antibody within the preceding 3 months. Prior treatment with live (attenuated) virus vaccine within the preceding 1 month.
* Patients taking hematopoietic cytokines within 2 weeks before enrollment.
* Patients with suspected active or latent TB infections.
* Patients with known active bacterial, viral, fungal, mycobacterium, parasitic or other infections (excluding fungal nail infection) or any serious systemic infections requiring intravenous antibiotic treatment or hospitalization (excluding neoplastic fever) in the 4 weeks prior to enrollment.
* Other serious conditions that may limit patients participation in the trial, such as Uncontrolled diabetes, Severe cardiac insufficiency (NYHA grade II or above), Acute coronary syndrome in the last 6 months, Coronary revascularization includes stent implantation, coronary artery bypass surgery, and other cardiac and vascular related procedures in the last 6 months, severe arrhythmia (including frequent ventricular premature beats, ventricular tachycardia , fast atrial fibrillation/ atrial flutter, severe bradycardia), Uncontrolled high blood pressure(>150/100mmHg), gastric ulcer(gastric ulcers were at risk of perforation), Active autoimmune disease, Severe hypertension, Severe respiratory disease(obstructive pulmonary disease or history of bronchospasm).
* Any contraindication of the CHOP drugs, including previously received anthracycline antibiotics; Patients with diabetes cannot tolerate prednisone therapy.
* Patients had a history of alcohol abuse or drug abuse.
* Allergic physique or known sensitivity or allergy to the active ingredient, excipient, murine products, heterologous proteins of any drug used in this treatment(including CHOP).
* Patients with serious mental illness.
* Patients who are unable to comply during the trial and/or follow-up phase.
* The researchers considered the patients unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-10 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Up to 3 years
  The complete response rate

SECONDARY OUTCOMES:
Progression-free survival | Up to 3 years
  PFS was defined as time from study registration to first disease progression or death whichever occurred first, otherwise subject data were censored at time last known disease free.
Overall Survival | Up to three years
  OS was defined as time from study registration to death, and otherwise censored at time last known alive.
Objective Remission Rate | Up to 2 years
  CR+PR

IPD SHARING:
Plan to Share IPD: Yes
YES